CLINICAL TRIAL: NCT02482662
Title: Assessment of the Diagnosis Test for Gestational Diabetes Mellitus
Brief Title: Diagnosis Test for Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-Luc Ardilouze, Endocinologist, Université de Sherbrooke
Other Study IDs: 14-159
Record Dates: First submitted 2015-06-16; First posted 2015-06-26 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Diagnosis
MeSH Terms: conditions — Diabetes, Gestational; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Diagnosis — Oral glucose tolerance test and self-monitoring blood glucose

SUMMARY:
Gestational diabetes mellitus (GDM) is an asymptomatic disease. Diagnosis is based on a oral glucose tolerance test (OGTT) requiring pregnant women to absorb 75g of glucose while fasting since midnight and to stay sober for another two hours. These OGTTs are poorly tolerated by pregnant women. As many OGTT are false positive according to self-monitoring blood glucose (SMBG), the investigators need now to determine the percentage of OGTT results that are false negative.

The comparison of the two tests (OGTT and SMBG) in the same patient with normal results of OGTT will determine the exact percentage of false negative OGTT results.

The opinion of women will also be taken into account. In the everyday clinic, many report that they prefer SMBG to OGTT because they do not have to be fasting, to drink non palatable drink and to attend a 2-hour visit in their schedule. However, no opinion study has yet been performed, the investigators will investigate formally what women think using a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* positive GDM screening test (glycemia post-50g of glucose ≥ 7.2 mmol/L),
* between 24 and 28 weeks of gestation from the last menstruation,
* single pregnancy,
* able to read and understand French.

Exclusion Criteria:

* known type 1 or type 2 diabetes,
* disease or treatment interfering with the metabolism of glucose,
* deficiency may hinder the understanding of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with abnormal GDM screening test.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
proportion of OGTTs falsely negative | Will be evaluated when participants finished SMBG i.e. 7 days after the OGTT

SECONDARY OUTCOMES:
preference of participants regarding the two tests (OGTT vs. SMBG) | Will be evaluated when participants finished SMBG i.e. 7 days after the OGTT
  Evaluated by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Ardilouze, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche clinique du CHUS, Sherbrooke, Quebec, Canada